CLINICAL TRIAL: NCT05297890
Title: A Phase 2, Multi-Center, Open-Label, Single-Arm Study to Evaluate the Efficacy and Safety of Lorlatinib Monotherapy in Crizotinib and Platinum-based Chemotherapy Treated Locally Advanced or Metastatic ROS1-Positive Non-Small Cell Lung Cancer Subjects in China
Brief Title: A Study of Lorlatinib in Subjects With ROS1-Positive Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS3011-201
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Advanced or Metastatic ROS1-Positive Non-Small Cell Lung Cancer
MeSH Terms: interventions — lorlatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lorlatinib (Experimental): Drug：Lorlatinib 100mg, oral, Quaque Die (QD), continuous administration in 21 days as a cycle
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — Dosage Form: Lorlatinib tablet, Dosage: 25mg/tablet, Dosing Regimens: 100mg, oral, Quaque Die (QD), continuous administration in 21 days as a cycle

SUMMARY:
A Phase 2, Multi-Center, Open-Label, Single-Arm Study to Evaluate the Efficacy and Safety of Lorlatinib Monotherapy in Crizotinib and Platinum-based Chemotherapy Treated Locally Advanced or Metastatic ROS1-Positive Non-Small Cell Lung Cancer (NSCLC)Subjects in China

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically or cytologically confirmed diagnosis of locally advanced or metastatic ROS1 gene arrangement positive NSCLC.
* Subject should have radiological disease progression while on treatment with crizotinib as the only prior ROS1 inhibitor.
* Participants must have been treated with platinum-based doublet chemotherapy for locally advanced/metastatic disease for at least 1 cycle and must have radiological disease progression on or after that. Participants who do not tolerate platinum-based doublet chemotherapy may be included provided they have been treated for at least 1 cycle.
* Prior treatment with small molecules or cytotoxic agents must have completed ≥5 half-lives prior to initiating study treatment; Prior treatment with antibodies must have completed at least 3 weeks prior to initiating study treatment.
* All Subjects must have at least 1 measurable target lesion (intracranial or extracranial) according to RECIST v1.1.
* Eastern Cooperative Oncology Group performance status (ECOG PS) 0, 1, or 2.
* Age ≥18 years.
* Subjects must have adequate organ function as assessed in the laboratory tests.
* Acute effects of prior anti-cancer treatment resolved to baseline severity or to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE 5.0) Grade 1 except for AEs that in the investigator's judgment do not constitute a safety risk for the subject.
* Serum or urine pregnancy test (for females of childbearing potential) negative at screening.
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
* Willing and able to comply with the study scheduled visits, treatment plans, laboratory tests, and other procedures.

Exclusion Criteria:

* More than 1 prior chemotherapy regimen prior to enrollment in the locally advanced/metastatic setting.
* Subject's cancer has a known primary driver alteration other than ROS1 gene rearrangement.
* Major surgery within 4 weeks prior to the first dose.
* Radiation therapy within 2 weeks prior to the first dose. Palliative radiation must have been completed at least 48 hours prior to the first dose. Stereotactic or partial brain irradiation must have completed at least 2 weeks prior to the first dose. Whole brain irradiation must have completed at least 4 weeks prior to the first dose.
* Spinal cord compression unless the subject has good pain control attained through therapy, and there is complete recovery of neurological function for the 4 weeks prior to the first dose.
* Gastrointestinal abnormalities, including inability to take oral medication; requirement for intravenous alimentation; prior surgical procedures affecting absorption including total gastric resection or lap band; active inflammatory gastrointestinal disease, chronic diarrhea, symptomatic diverticular disease; treatment for active peptic ulcer disease in the past 6 months; malabsorption syndromes.
* Known prior or suspected severe hypersensitivity to lorlatinib or any component in the formulation; known prior therapy with lorlatinib.
* Severe acute or chronic infections.
* Clinically significant cardiovascular disease (both arterial and venous) and non-vascular cardiac conditions (active or within 3 months prior to the first dose).
* Subject with predisposing characteristics for acute pancreatitis according to investigator judgment, including but not limited to uncontrolled hyperglycemia, current gallstone disease, in the last month prior to the first dose.
* History of extensive, disseminated, bilateral or presence of Grade 3 or 4 interstitial fibrosis or interstitial lung disease including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis and pulmonary fibrosis.
* Evidence of active malignancy within the last 3 years prior to the first dose.
* Concurrent use of any of the prohibited food or drugs required in protocol within 12 days prior to the first dose of administration of lorlatinib.
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, would make the subject inappropriate for entry into this study.
* Participation in other studies involving investigational drug(s) within 2 weeks prior to study entry and/or during study participation.
* Pregnant female subjects; breastfeeding female subjects.
* Any use of traditional Chinese medicines or herbal preparations with anti-tumor indications within 7 days before the first dose of investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 per Independent Central Radiology (ICR) assessment | From the date of first dose of first subject to 6 months after the first dose of last subject, assessed up to approximately 19 months

SECONDARY OUTCOMES:
Duration of response (DoR) as assessed by RECIST v1.1 per ICR assessment | From the date of first dose of first subject to 6 months after the first dose of last subject, assessed up to approximately 19 months
ORR assessed by RECIST version 1.1 per investigator assessment | From the date of first dose of first subject to 6 months after the first dose of last subject, assessed up to approximately 19 months
DoR assessed by RECIST version 1.1 per investigator assessment | From the date of first dose of first subject to 6 months after the first dose of last subject, assessed up to approximately 19 months
Disease control rate (DCR) at 12 and 24 week as assessed by RECIST v1.1 per ICR assessment | From the date of first dose of first subject to 6 months after the first dose of last subject, assessed up to approximately 19 months
Time to tumor response (TTR) as assessed by RECIST v1.1 per ICR assessment | From the date of first dose of first subject to 6 months after the first dose of last subject, assessed up to approximately 19 months
Progression-free survival (PFS) as assessed by RECIST v1.1 per ICR assessment | From the date of first dose of first subject to 6 months after the first dose of last subject, assessed up to approximately 19 months
Intracranial Objective Response (IC-OR) as assessed by RECIST v1.1 per ICR assessment | From the date of first dose of first subject to 6 months after the first dose of last subject, assessed up to approximately 19 months
Duration of intracranial response (IC-DoR) as assessed by RECIST v1.1 per ICR assessment | From the date of first dose of first subject to 6 months after the first dose of last subject, assessed up to approximately 19 months
Overall survival (OS) | From the date of first dose of first subject to 6 months after the first dose of last subject, assessed up to approximately 19 months
To evaluate the safety and tolerability of lorlatinib treatment | From the date of first dose of first subject to 6 months after the first dose of last subject, assessed up to approximately 19 months
Lorlatinib concentration will be used for population PK analysis | From the date of first dose of first subject to 6 months after the first dose of last subject, assessed up to approximately 19 months
patient-reported outcomes (PROs) as assessed by EORTC QLQ-C30 and EORTC QLQ-LC13 (self-assessment questionnaires) | From the date of first dose of first subject to 6 months after the first dose of last subject, assessed up to approximately 19 months

CONTACTS AND LOCATIONS:
Locations (31):
- China (31):
  - Guangdong Provincial People's hospital, Guangzhou, Guangdong
  - Beijing Cancer Hospital, Beijing
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - The First Hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - Sichuan Cancer Hospital & Institute, Chengdu
  - West China Hospital of Sichuan University, Chengdu
  - Chinese PLA Army Medical Center, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - The first Affiliated hospital, Sun Yat-Sen University, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Shandong Cancer Hospital&Institute, Jinan
  - Yunnan Cancer Hospital, Kunming
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu Province Hospital, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Liaoning Cancer Hospital and Institute, Shenyang
  - Shanxi Cancer hospital, Taiyuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - The 1st Affiliated hospital of Wenzhou Medical University, Wenzhou
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Tangdu Hospital of The fourth Military Medical University Peoples Liberation Army of China, Xi'an
  - Xiamen Humanity Hospital, Xiamen
  - Henan Cancer Hospital, Zhengzhou
  - Henan Provincial People's Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou